CLINICAL TRIAL: NCT05356182
Title: A Pilot and Feasibility Study of a Dietary Intervention With Low-protein Meals in Cancer Patients Receiving Immunotherapies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Roberto Pili, Associate Dean for Cancer Research and Integrative Oncology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005755
Record Dates: First submitted 2022-04-01; First posted 2022-05-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Medical Oncology; Integrative Oncology; Medical Nutrition Therapy
Keywords: Oncology; Nutrition; Immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Diet Arm (Active Comparator): control diet arm (~20% protein content)
  Interventions: Other: Diet
- Low-Protein Diet Arm (Active Comparator): intervention low-protein diet arm (10% protein content)
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Control diet consisting of 20% protein, intervention diet consisting of 10% protein

SUMMARY:
The main idea of this study is that a low protein diet may alter the environment surrounding the tumor, enhancing the body's immune response leading to greater anticancer effects of treatment. This study intends to use a low-protein diet as a tool to enhance the immune response generated by immune check point inhibitor treatments.

DETAILED DESCRIPTION:
This is a single center, randomized, open label study to assess the feasibility of a low-protein diet intervention in cancer patients who are receiving immunotherapies. Subjects will be randomized in a 1:1 ratio to either immunotherapy plus control diet arm (~20% protein content) or immunotherapy plus intervention low-protein diet arm (10% protein content).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented solid tumor malignancies which is amenable for immunotherapy treatment with immune checkpoint inhibitors (i.e. PD1, PD-L1, CTLA inhibitors) as single agents or in combination.
* Metastatic disease as evidenced by soft tissue and/or bony metastases on baseline bone scan and/or computed tomography (CT) scan of the chest, abdomen, and pelvis
* Life expectancy of at least 6 months
* Adults ≥ 18 years of age
* Adequate hematologic, renal, and liver function as evidenced by the following:

  * White blood cell (WBC) ≥ 2,500 cells/μL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/μL
  * Platelet Count ≥ 100,000 cells/μL
  * Hemoglobin (HgB) ≥ 9.0 g/dL
  * Creatinine ≤ 2.0 mg/dL
  * Total bilirubin ≤ 2 x upper limit of normal (ULN)
  * Aspartate aminotransaminase (AST, SGOT) ≤ 2.5 x ULN
  * Alanine aminotransaminase (ALT, SGPT) ≤ 2.5 x ULN

Exclusion Criteria:

* • Eastern Cooperative Oncology Group (ECOG) performance status 2 or higher

  * Treatment with any of the following medications or interventions within 28 days of registration:

    * Systemic corticosteroids; however, use of inhaled, intranasal, and topical steroids is acceptable.
    * High dose calcitriol [1,25(OH)2VitD] (i.e., > 7.0 μg/week)
  * A requirement for systemic immunosuppressive therapy for any reason
  * Any infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5°F or 38.1°C) within 1 week prior to registration
  * A known allergy, intolerance, or medical contraindication to receiving the contrast dye required for the protocol-specified CT imaging
  * Any medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of low-protein diet intervention in cancer patients receiving immunotherapies. | 4 Months
  Change in blood urea nitrogen (BUN) from baseline to post-intervention (following 3 cycles of treatment) will be measured to assess adherence of following the diet intervention.
To assess the feasibility of low-protein diet intervention in cancer patients receiving immunotherapies. | 4 Months
  Change in urine urea nitrogen (UUN) from baseline to post-intervention (following 3 cycles of treatment) will be measured to assess adherence of following the diet intervention.

SECONDARY OUTCOMES:
To assess whether low-protein diet intervention augments the immune response to immunotherapies in cancer patients receiving immunotherapies | 4 Months
  Includes isolation and characterization of antigen specific T cell clones
To assess whether low-protein diet intervention augments the immune response to immunotherapies in cancer patients receiving immunotherapies | 4 Months
  Includes evaluation of antigen specific T cell populations by spectratyping T cell receptor expression
To assess whether low-protein diet intervention augments the immune response to immunotherapies in cancer patients receiving immunotherapies | 4 Months
  Includes characterization of antigen response by cytokine and chemokine production
To assess the enrollment rate (safety and tolerability) of the combination of immunotherapies and low-protein diet intervention | 4 Months
  Enrollment rate
To assess the Drop-out rate (safety and tolerability) of the combination of immunotherapies and low-protein diet intervention | 4 Months
  Drop-out rate
To assess the safety and tolerability of the combination of immunotherapies and low-protein diet intervention | 4 Months
  Compliance with diet measured by self-report of patient
To obtain preliminary evidence of clinical efficacy of immunotherapies and low-protein diet compared to immunotherapies and control-diet using the RECIST v1.1 criteria | 4 Months
  Objective Response Rate (ORR)
To obtain preliminary evidence of clinical efficacy of immunotherapies and low-protein diet compared to immunotherapies and control-diet using the RECIST v1.1 criteria | 4 Months
  Progression-Free Survival (PFS)
To obtain preliminary evidence of clinical efficacy of immunotherapies and low-protein diet compared to immunotherapies and control-diet using the RECIST v1.1 criteria | 4 Months
  Overall Survival(OS)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo / Great Lakes Cancer Care, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided